CLINICAL TRIAL: NCT07167303
Title: The Effect of Scenario-Based Gamified Virtual Reality Application on Nurses' Knowledge Level in Basic Life Support Practices: A Randomized Controlled Trial
Brief Title: Virtual Reality Application in Basic Life Support Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Duygu Akbas Uysal, Principal Investigator Dr, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1919
Record Dates: First submitted 2025-08-26; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Cardiopulmonary Resuscitation (CPR); Nursing Education Research; Virtual Reality; Randomized Controlled Trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (VR Training): (Experimental): Participants were first introduced to the VR simulator and briefed on the current scenario. Through the VR headset, nurses experienced the CPR scenario in real time in an interactive environment. Each nurse had sufficient time to practice the skill steps in the given scenario. Participants used the scenario-based VR CPR training game until they felt ready (approximately 30 minutes)
  Interventions: Other: VR Training)
- Control Group (Traditional Training) (Active Comparator): Nurses in the control group received traditional training in a hospital training room using an adult plastic CPR manikin (approximately 30 minutes).
  Interventions: Other: Traditional Training

INTERVENTIONS:
Other: VR Training) — Participants were first introduced to the VR simulator and briefed on the current scenario. Through the VR headset, nurses experienced the CPR scenario in real time in an interactive environment. Each nurse had sufficient time to practice the skill steps in the given scenario. Participants used the scenario-based VR CPR training game until they felt ready (approximately 30 minutes)
  Arms: Intervention Group (VR Training):
Other: Traditional Training — Nurses in the control group received traditional training in a hospital training room using an adult plastic CPR manikin
  Arms: Control Group (Traditional Training)

SUMMARY:
Introduction: This study investigates the effect of virtual reality (VR)-based training methods on the acquisition of cardiopulmonary resuscitation (CPR) skills and user attitudes within the framework of Kolb's Experiential Learning Model.

Methods: A randomized controlled trial was conducted between December 11, 2024, and August 11, 2025, with 60 nurses (30 in the experimental group and 30 in the control group) working in emergency and intensive care units. The experimental group practiced an interactive CPR scenario using VR headsets, while the control group received CPR training through traditional methods. Data were collected using a descriptive information form, a knowledge test, and the Virtual Reality Attitude Scale. The knowledge test, prepared in accordance with the American Heart Association (AHA) standards, was administered as a pre-test, post-test, and follow-up test two weeks later. Additionally, the VR Satisfaction Scale was applied to the experimental group.

ELIGIBILITY:
Inclusion Criteria:

Ability to use virtual reality (VR) glasses Being an emergency room nurse or an intensive care nurse

Exclusion Criteria:

Having difficulty in communication

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-12-11 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-08-11 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure Change in knowledge scores on Basic Life Support - Description: Knowledge level will be assessed using a BLS knowledge test prepared in accordance with American Heart Association standards. Sub-dimensions include Airwa | Pre-test (baseline), Post-test (immediately after intervention), and Two-week follow-up.
  The 18-question form assesses five different competency areas: Basic Life Support, Airway and Breathing, Chest Compressions, Automatic External Defibrillator Use, and Communication with Continuity of CPR. For each question, nurses selected either "True" or "False," with a correct answer receiving 1 point and an incorrect answer receiving 0 points. The highest score is 18, and the lowest is 0.A higher score indicates a higher level of knowledge.

SECONDARY OUTCOMES:
Secondary Outcomes Virtual Reality Attitude Scale - Measurement of participants' attitudes toward VR-based training. - Correlation between VR attitude scores and knowledge test scores (e.g., post-test and pre-post difference scores). | At baseline (pre-intervention), immediately post-intervention, and at 2 weeks follow-up
  1. Virtual Reality Attitude Scale
  * Measurement of participants' attitudes toward VR-based training.
  * Correlation between Virtual Reality Attitude Scale attitude scores and knowledge test scores (e.g., post-test and pre-post difference scores).
  Possible scores range from 9 to 45, and there are no reverse items. A higher score indicates a stronger attitude toward virtual reality.

CONTACTS AND LOCATIONS:
Locations (1):
- Tinaztepe Universty, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No